CLINICAL TRIAL: NCT02089477
Title: The Smart-phone as a Physical Fitness Monitor on a Population Level - Validity and Sensitivity and Improtance of Individual Motivation for Doing Interval Walking With the InterWalk Application
Brief Title: The Smart-phone as a Physical Fitness Monitor - Validity, Sensitivity and Motivation InterWalk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Staun Valentiner (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Laura Staun Valentiner, PhD-student, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: InterWalk - Validation
Record Dates: First submitted 2014-03-14; First posted 2014-03-17 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes, InterWalk, Individual Support, Motivation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Support (Experimental): The participants in the intervention group receives the intervention and support consisting of:
  1. Individual Goal Setting: 2-3 functional goals related to everyday life evaluated every 4th week.
  2. SMS send every Sunday with 5 possible responses. depending on the answer of the participant it will cause a telephone call from a project about motivation and barriers for interval walking.
  Interventions: Other: Support group
- Control group (No Intervention): Patient's in the control group receives the intervention with interval Walking and no other support.

INTERVENTIONS:
Other: Support group — The participants in the intervention group receives the intervention and support consisting of:
  1. Individual Goal Setting: 2-3 functional goals related to everyday life evaluated every 4th week.
  2. SMS send every Sunday with 5 possible responses. depending on the answer of the participant it will cause a telephone call from a project about motivation and barriers for interval walking.
  Arms: Support

SUMMARY:
Low physical fitness may cause several life style related diseases e.g. cardiovascular disease, cancer and type 2 diabetes. It is important to develop reliable methods for measurement which can be used to follow the development of the physical shape both on an individual level and on at population level.

Associated with the development of new training method known as Interval Walking we developed an application for smartphones. The use of the application InterWalk was meant to increase physical activity in patients with type 2 diabetes. The application should both be able to, 1) be a personal trainer when doing interval walking, and 2) measure the individual physical fitness performed as a walking test. The latter function was developed to make the training more personal and individal adapted, so that the training was neither too hard or too easy.

It is necessary to test the walking test against a golden standard for measuring physical fitness and that the test in the application is able to measure and register changes in physical fitness.

Our hypothesis is that the individual test, in the InterWalk Application is reliable and able to register changes in physical fitness in patients with type 2 diabetes. The purpose of this project is investigate the reliability of a smartphone-based test of physical fitness, and to investigate whether the test is able to register changes in physical fitness during the project time (3 month). A secondary aim is to investigate whether individual support during the training period, affect the individual effort and time of interval walking per week.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, age 30-80 y, BMI >18 but <40 kg/m2 and confirmed T2D diagnose

Exclusion Criteria:

* Pregnancy, smoking, contraindication to increased levels of physical activity, insulin dependence, evidence of thyroid, liver, lung, heart or kidney disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome is amount of time duing interval walking (in minuts) with InterWalk per week after 3 month | up to 3 months after enrollment

SECONDARY OUTCOMES:
Frequency of Interval walking with InterWalk | 3 months after enrollment
Quality of data with VO2-peek test in the InterWalk Application | 3 months after enrollment
  quantity of minuts with high and low intervals after 3 month
validation of InterWalk, VO2-peek test | 3 months after enrollment
VO2-peek test in the InterWalk Application | 3 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Ried-Larsen, Post Doc, Principal Investigator — CIM, University Hospital Rigshospitalet
Locations (1):
- Center of Inflammation and Metabolism, Copenhagen, Denmark

REFERENCES:
- [Derived] Valentiner LS, Thorsen IK, Kongstad MB, Brinklov CF, Larsen RT, Karstoft K, Nielsen JS, Pedersen BK, Langberg H, Ried-Larsen M. Effect of ecological momentary assessment, goal-setting and personalized phone-calls on adherence to interval walking training using the InterWalk application among patients with type 2 diabetes-A pilot randomized controlled trial. PLoS One. 2019 Jan 10;14(1):e0208181. doi: 10.1371/journal.pone.0208181. eCollection 2019. PMID 30629601
- [Derived] Karstoft K, Brinklov CF, Thorsen IK, Nielsen JS, Ried-Larsen M. Resting Metabolic Rate Does Not Change in Response to Different Types of Training in Subjects with Type 2 Diabetes. Front Endocrinol (Lausanne). 2017 Jun 13;8:132. doi: 10.3389/fendo.2017.00132. eCollection 2017. PMID 28659869
- [Derived] Brinklov CF, Thorsen IK, Karstoft K, Brons C, Valentiner L, Langberg H, Vaag AA, Nielsen JS, Pedersen BK, Ried-Larsen M. Criterion validity and reliability of a smartphone delivered sub-maximal fitness test for people with type 2 diabetes. BMC Sports Sci Med Rehabil. 2016 Oct 7;8:31. doi: 10.1186/s13102-016-0056-7. eCollection 2016. PMID 28174664